CLINICAL TRIAL: NCT04365660
Title: A Phase 2 Study of 18F FTC 146 PET/CT in Patients With Newly Diagnosed Osteosarcoma
Brief Title: 18F-FTC-146 PET/CT in Newly-Diagnosed Osteosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual with no intent of continuing
Sponsor: Davidzon, Guido, M.D. (Other)
Responsible Party: Principal Investigator, Kristen Ganjoo, Professor of Medicine (Oncology), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-52746; SARCOMA0041 (Other: OnCore); IRB-52746 (Other: Stanford IRB); NCI-2021-03443 (Registry Identifier: CTRP)
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18-F-FTC 146 PET/CT (Experimental): For PET scans, subjects will receive intravenous injection of 10 mCi 18-F -FTC 146 administered twice with 18-F-FTC 146, once at baseline (pre chemotherapy) and once at final study visit (post chemotherapy).
  Interventions: Drug: 18-F FTC 146

INTERVENTIONS:
Drug: 18-F FTC 146 — Radiotracer, 10 mCi at pre- and post- chemotherapy, intravenous administration

SUMMARY:
The purpose of this research is to evaluate the study drug, 18F FTC-146, as a positron emission tomography (PET) / computed tomography (CT) radiotracer imaging agent to evaluate tumor status in patients newly diagnosed with osteosarcoma ("bone cancer").

DETAILED DESCRIPTION:
Primary Objective: Demonstrate correlation of pre-post reduction in 18F-FTC-146 PET/CT with amount of post-treatment tumor necrosis in newly-diagnosed and treated osteosarcoma patients.

Secondary Objective: Demonstrate correlation of pre-post reduction in 18F-FTC-146 PET/CT with amount of post-treatment pain reduction in newly-diagnosed and treated osteosarcoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven osteosarcoma requiring local surgical intervention.
* ECOG ≤ 2
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Chemotherapy in the past 2 months.
* Prior history of allergic reaction to 18F FTC 146.
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen N Ganjoo, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 18-F-FTC 146 PET/CT: For PET scans, intravenous injection of 10 mCi 18-F -FTC 146 administered twice with 18-F-FTC 146, once at baseline (pre chemotherapy) and once at final study visit (post chemotherapy).
Period: Overall Study
Arm/Group | 18-F-FTC 146 PET/CT
Started | 1
Received PET/CT Scan | 0
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | 18-F-FTC 146 PET/CT
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Detection of Tumor Necrosis Post-chemotherapy
Description: Participants will be assessed with 18F FTC 146 PET/CT imaging at baseline and after neoadjuvant (pre surgery) chemotherapy but before surgery itself. Chemotherapy will be nominally three 3 week cycles administered over up to 12 weeks. The ability of 18F FTC 146 PET/CT to evaluate treatment effect will be assessed as the percentage of tumor that is assessed as necrotic after the treatment course. The outcome will be reported as the mean percentage of the resected tumor (removed by surgery) that is assessed by histopathology as necrotic, with standard deviation.
Time Frame: 12 weeks
Population: No data were collected for this outcome measure.
Arm/Group | 18-F-FTC 146 PET/CT
Number analyzed (Participants) | 0

2. Secondary Outcome: Maximum Standardized Uptake Value (SUVmax)
Description: Participants will be assessed with 18F FTC 146 PET/CT imaging at baseline and after neoadjuvant (pre surgery) chemotherapy but before surgery itself. Chemotherapy will be nominally three 3 week cycles administered over up to 12 weeks. Based on the PET/CT scans, the maximum standardized uptake value (SUVmax) in the tumor region of interest (ROI) will be calculated at baseline and after treatment. The outcome will be reported as the mean percent change in SUVmax from baseline to post treatment, with standard deviation.
Time Frame: 12 weeks
Population: No data were collected for this outcome measure.
Arm/Group | 18-F-FTC 146 PET/CT
Number analyzed (Participants) | 0

3. Secondary Outcome: Use of Patient Reported Outcomes Measurement Information System (PROMIS) to Assess Treatment Effect
Description: Participants will receive neoadjuvant (pre surgery) chemotherapy, nominally three 3 week cycles administered over up to 12 weeks. The treatment effect of the neoadjuvant chemotherapy will be assessed as the change in scores on the PROMIS (Patient Reported Outcomes Measurement Information System) questionnaire, from baseline to post treatment. The result will be reported as the mean difference from baseline to post treatment, with standard deviation.
Time Frame: 12 weeks
Population: No data were collected for this outcome measure.
Arm/Group | 18-F-FTC 146 PET/CT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | 18-F-FTC 146 PET/CT
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04365660/Prot_SAP_001.pdf